CLINICAL TRIAL: NCT03571646
Title: LIFEGUARD Study - Continuous Respiratory Monitoring on the General Ward
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment rate due to difficulties in identifying suitable patients
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: MDT17026
Record Dates: First submitted 2018-05-02; First posted 2018-06-27 (Actual); Results first posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Respiratory Complication

STUDY DESIGN:
Intervention Model Description: The occurrence of at least one of the following RC markers will be considered as primary endpoint for patients monitored by Capnostream 20p during both study Phases: (1) SpO2 ≤ 90% for ≥ 3 minutes.(2) RR ≤ 8 or ≥ 22 bpm for ≥ 3 minutes. (3) etCO2 ≤ 15 or ≥ 60 mmHg for ≥ 3 minutes. (4) Apnea episode lasting > 30 seconds.
  The occurrence of at least one of the following RC markers will be considered as primary endpoint for patients monitored by PM1000N-RR during both study Phases:
  (1) SpO2 ≤ 90% for ≥ 3 minutes. (2) RR ≤ 8 or ≥ 22 bpm for ≥ 3 minutes.
Who Masked: Care Provider
Masking Description: During the study Phase I, the alarms of both devices will be silenced and the screen information blinded, as is the current clinical practice. During the study Phase II, the screen information will be available and the nursing staff will be instructed to respond to both devices' alarms based on a pre-defined hospital protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Capnostream 20 (Other): Continuous monitoring of CO2
  Interventions: Behavioral: Capnostream 20 monitoring
- PM1000N-RR (Other): Continuous monitoring of SpO2
  Interventions: Device: PM1000N-RR monitoring

INTERVENTIONS:
Behavioral: Capnostream 20 monitoring — Continuous monitoring on a general ward
  Arms: Capnostream 20
Device: PM1000N-RR monitoring — Continuous monitoring on a general ward
  Arms: PM1000N-RR

SUMMARY:
The purpose of this study is to document how often and how severe are the breathing difficulties that patients suffer, while recovering on a general ward following a serious operation

DETAILED DESCRIPTION:
This is a prospective, 2-center, 2-phase pilot study of post-surgical adult patients on the hospital ward at high risk of developing respiratory and cardiovascular events. Phase I, 70 patients will be 1:1 randomly allocated to Capnostream 20p monitoring system or to PM1000N-RR pulse oximeter monitoring system and the alarms of both devices will be silenced and the screen information blinded, to establish a baseline for the incidence of respiratory events. Phase II, 140 patients will be 1:1 randomly allocated to Capnostream 20p or to PM1000N-RR monitoring but the screen information will be visible at the bedside and through the Vital Sync™ remote patient monitoring system.

ELIGIBILITY:
Inclusion Criteria:

* Non-cardiac post-surgical patients at high risk of developing respiratory and cardiovascular events (High or intermediate risk for postoperative pulmonary complications).
* Adult age (≥18 year old).
* Patient is able and willing to give informed consent.

Exclusion Criteria:

* Expected ward length of stay ≤24 hours.
* Post-surgical patients with American Society of Anesthesiologists physical status (ASA PS) V or higher.
* Ventilated or intubated patients.
* Patient is unwilling or unable to comply fully with study procedures due to any disease condition which can raise doubt about compliance
* Patient is a member of a vulnerable population regardless of authorized representative support.
* Patient is participating in another potentially confounding drug or device clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2019-12-14 (Actual); Study Completion 2019-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Hoeft, MDPhD, Principal Investigator — Universitätsklinikum Bonn (AöR), D-53127 Bonn - Germany; Michael Sander, Dr.Med, Principal Investigator — Universitätsklinikum Gießen und Marburg (UKGM) , 20043 Marburg - Germany
Locations (2):
- Germany (2):
  - Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Gießen und Marburg, Marburg

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Capnostream 20 | PM1000N-RR
Started | 3 | 3
Completed | 1 | 2
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Capnostream 20 | PM1000N-RR | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Customized [Mean (Standard Deviation); unit: years] | NA (NA) — data analysis was not performed due to the early termination of the study | NA (NA) — data analysis was not performed due to the early termination of the study | NA (NA) — data analysis was not performed due to the early termination of the study
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — data analysis was not performed due to the early termination of the study | NA — data analysis was not performed due to the early termination of the study | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — data analysis was not performed due to the early termination of the study | NA — data analysis was not performed due to the early termination of the study | NA — Total not calculated because data are not available (NA) in one or more arms.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | NA — data analysis was not performed due to the early termination of the study | NA — data analysis was not performed due to the early termination of the study | NA — Total not calculated because data are not available (NA) in one or more arms.
Height [Mean (Standard Deviation); unit: cm] | NA (NA) — data analysis was not performed for this study due to early termination and insufficient data collection | NA (NA) — data analysis was not performed for this study due to early termination and insufficient data collection | NA (NA) — data analysis was not performed for this study due to early termination and insufficient data collection
weight [Mean (Standard Deviation); unit: kg] | NA (NA) — data analysis was not performed for this study due to early termination and insufficient data collection | NA (NA) — data analysis was not performed for this study due to early termination and insufficient data collection | NA (NA) — data analysis was not performed for this study due to early termination and insufficient data collection
shirt collar neck size [Mean (Standard Deviation); unit: cm] | NA (NA) — data analysis was not performed for this study due to early termination and insufficient data collection | NA (NA) — data analysis was not performed for this study due to early termination and insufficient data collection | NA (NA) — data analysis was not performed for this study due to early termination and insufficient data collection
at what elevation does subject reside [Mean (Standard Deviation); unit: METERS] | NA (NA) — data analysis was not performed for this study due to early termination and insufficient data collection | NA (NA) — data analysis was not performed for this study due to early termination and insufficient data collection | NA (NA) — data analysis was not performed for this study due to early termination and insufficient data collection
ARISCAT score [Mean (Standard Deviation); unit: units on a scale] — ARISCAT Score is an accurate risk score for predicting high or intermediate risk for postoperative pulmonary complications in patients undergoing surgery, calculated based on preoperative data such as on patient's age, preoperative SpO2, respiratory infection, anemia, surgery type and duration.
  An ARISCAT score of ≥ 26 indicates high or intermediate risk for postoperative pulmonary complications.
  Low risk: <26, Intermediate risk: 26-44, High risk: ≥45 No theoretical minimum and maximum score exists; scores are calculated based on patient variables (listed above).
  units on a scale | NA (NA) — data analysis was not performed for this study due to early termination and insufficient data collection | NA (NA) — data analysis was not performed for this study due to early termination and insufficient data collection | NA (NA) — data analysis was not performed for this study due to early termination and insufficient data collection
POSPOM score [Mean (Standard Deviation); unit: units on a scale] — POSPOM Score is an accurate risk score for predicting in-hospital mortality in patients undergoing surgery, calculated based on preoperative data such as on patient's age, planned surgery and presence of additional diseases or disorders.
  POSPOM <20: Average risk (less than 0.4% predicted risk) POSPOM=24: 3 times the average risk (1.2%) POSPOM=28: 10 times the average risk (4.2%) POSPOM=33: 40 times the average risk (16.5%) No theoretical minimum and maximum score exists as scores are calculated based on patient variables (listed above).
  units on a scale | NA (NA) — data analysis was not performed for this study due to early termination and insufficient data collection | NA (NA) — data analysis was not performed for this study due to early termination and insufficient data collection | NA (NA) — data analysis was not performed for this study due to early termination and insufficient data collection

OUTCOME MEASURES:

1. Primary Outcome: Quantify the Incidence and Severity of Post-operative Respiratory Compromise Markers
Description: Respiratory Compromise markers are identified by continuous monitoring to determine the benefit of continuous monitoring on the general ward
Time Frame: 72 hours
Population: Study was stopped prematurely due to difficulties with enrollment and low participation rate. A decision was made not to analyze data as only 6 patients were enrolled which would not give meaningful results.
Arm/Group | Capnostream 20 | PM1000N-RR
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Evaluate 2 Different Monitoring Devices
Description: Compare patient compliance and the sensitivity of two monitoring systems in high risk, post-surgical patients Study was stopped prematurely due to difficulties with enrollment and low participation rate. A decision was made not to analyze data as only 6 patients were enrolled which would not give meaningful results.
Time Frame: 72 hours
Population: as for outcome 1
Arm/Group | Capnostream 20 | PM1000N-RR
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Capnostream 20 | PM1000N-RR
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 1/3 | 0/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Capnostream 20 (N=3) | PM1000N-RR (N=3)
transfer back to intermediate care (IMC) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — AFTER PATIENT RETURNED FROM IMC TO NORMAL WARD, SHE BECAME WORSE WITH HER LUNGS. THE LETTER TO THE DR DESCRIBES POSTOPERATIVE PLEURAL EFFUSION ON BOTH SIDES.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-06-19): https://cdn.clinicaltrials.gov/large-docs/46/NCT03571646/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-19): https://cdn.clinicaltrials.gov/large-docs/46/NCT03571646/SAP_001.pdf